CLINICAL TRIAL: NCT00895999
Title: Psychosocial Treatment for Gynecology Patients With Comorbid Depression and Pain
Brief Title: Psychosocial Treatment for Women With Depression and Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Ellen Poleshuck, Assistant Professor, Department of Psychiatry, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Poleshuck K23; 5K23MH079347 (NIH)
Record Dates: First submitted 2009-05-08; First posted 2009-05-11 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-03

CONDITIONS: Pelvic Pain; Depression
MeSH Terms: conditions — Pelvic Pain; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Female patients (n=30) who meet criteria for major depression and chronic pelvic pain will be randomly assigned to 8 individual sessions of IPT adapted for depression and pain.
  Interventions: Behavioral: Interpersonal Therapy for Pain (IPT-P)
- 2 (Other): Female patients (n=30) who meet criteria for major depression and chronic pelvic pain will be randomly assigned to Enhanced Support and Connection to Counseling (ESCC).
  Interventions: Behavioral: Enhanced Support and Connection to Counseling

INTERVENTIONS:
Behavioral: Interpersonal Therapy for Pain (IPT-P) — IPT-P focuses on improving relationships as a way to improve depression and pain. The patient and therapist work together to improve communication and enhance relationships and social support. Patients choose a problem focus and goal related to both their pain and depression. Up to 8 IPT-P sessions are provided regardless of ability to pay.
  Arms: 1
Behavioral: Enhanced Support and Connection to Counseling — Research staff connect patients with the Strong Family Therapy Services, Women's Behavioral Health Service, or other appropriate mental health care and reduce potential barriers from making it to the initial appointment. This support includes navigating insurance issues, addressing issues of childcare and transportation, helping to schedule the initial appointment, reminder calls, and follow-up after the scheduled intake. Research staff will also check-in monthly to see if the patients require any additional support to remain in mental health treatment. Up to 8 therapy sessions are covered regardless of ability to pay.
  Arms: 2

SUMMARY:
Patients with depression and pain have poorer outcomes in response to depression treatments than depressed patients without pain. While psychotherapy treatment studies have demonstrated improvement in pain and depression, no psychosocial interventions have been developed and tested prospectively specifically for patients with both conditions. Interpersonal psychotherapy (IPT), an effective treatment for depression, has been adapted successfully for physically ill patients and demonstrates good adherence, treatment satisfaction, and depression outcomes. The investigators propose to test a modified form of IPT-P for depressed patients with co-morbid pain.

ELIGIBILITY:
Inclusion Criteria:

* major depression
* chronic pelvic pain

Exclusion Criteria:

* current or past psychosis
* moderate mental retardation or greater
* active suicidal intent
* active abuse of non-prescribed substances (< 3 months)
* current individual psychotherapy
* current pregnancy
* terminal illness
* inability to communicate in English
* men

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2007-03; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
A self-report measure BDI and a clinician measure HRSD will evaluate depression severity. These measures are standards in primary care depression trials and in pain studies and have demonstrated sensitivity to detect changes in depress | 0, 12 wks, 24 wks, 36 wks

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Poleshuck, PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

REFERENCES:
- [Derived] Poleshuck E, Wittink M, Crean H, Gellasch T, Sandler M, Bell E, Juskiewicz I, Cerulli C. Using patient engagement in the design and rationale of a trial for women with depression in obstetrics and gynecology practices. Contemp Clin Trials. 2015 Jul;43:83-92. doi: 10.1016/j.cct.2015.04.010. Epub 2015 Apr 30. PMID 25937505
- [Derived] Poleshuck EL, Gamble SA, Bellenger K, Lu N, Tu X, Sorensen S, Giles DE, Talbot NL. Randomized controlled trial of interpersonal psychotherapy versus enhanced treatment as usual for women with co-occurring depression and pelvic pain. J Psychosom Res. 2014 Oct;77(4):264-72. doi: 10.1016/j.jpsychores.2014.07.016. Epub 2014 Jul 26. PMID 25280823